CLINICAL TRIAL: NCT04756011
Title: Aspects of Diabetes Technology (Insulin Pumps) Children Perspective, a Cross - Sectional Study
Brief Title: Health-related Quality of Life and Psychosocial Aspects of Diabetes Technology (Insulin Pumps)
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: Health related quality of life
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: T1DM; Health Related Quality of Life; Insulin Pump
Keywords: Insulin pump; T1DM; HRQL
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 11 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (insulin pump): 30 patients who are on insulin pump.
  Interventions: Other: Health related quality of life
- Group B (MDI): 30 patients who are on multiple daily injection.
  Interventions: Other: Health related quality of life

INTERVENTIONS:
Other: Health related quality of life — Confidence in diabetes self care questionnaire the socioeconomic level of the family scale MINI-KID the Peds-QL

SUMMARY:
This study will be prospective comparative trial comparing between insulin pumps vs Multiple daily injections (MDI) in treatment of type 1 diabetes mellitus (T1DM) in terms of health- related quality of life (HRQL) and efficacy of glycemic control (HbA1c level )

Hypothesis:

Type 1 diabetes is characterized by autoimmune destruction of insulin-secreting pancreatic b cells leading to disturbed glucose regulation and overt hyperglycemia which leads to variable consequences and complication. Consequently, individuals with type 1 diabetes have a lifelong dependency on insulin replacement therapy.

Aim of the Work:

To compare the psychosocial impact of insulin pumps versus multiple daily injections in treatment of type 1 diabetes mellitus (Via questionnaire) in terms of health-related quality of life and efficacy of glycemic control (HbA1c level).

ELIGIBILITY:
Inclusion Criteria:

* 1.Type 1 diabetes mellitus.
* 2.Patients who are on insulin pumps must be for at least 3 months on them

Exclusion Criteria:

* 1. Other types of DM e.g., T2DM, MODY.
* 2. Patients with other comorbidities; cardiac, renal, neurological, hepatic ….etc.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from Ain shams pediatric and adolescent diabetes unit(PADU)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Confidence in diabetes self care questionnaire (CIDS) | 10 min
  the CIDS scale, assessment included HbA1c, emotional distress, fear of hypoglycemia, self-esteem, anxiety, depression, and self-care behavior. The CIDS scale is a reliable and valid measure of diabetes-specific self-efficacy for use in patients with type 1 diabetes. High psychometric similarity allows for cross-cultural comparisons.
socioeconomic level of the family scale | 5 minutes
  Assessment of family socioeconomic standard
MINI-KID (Mini International Neuropsychiatric Interview ) | 25 minutes
  Mini International Neuropsychiatric Interview for Children and Adolescents
Evaluation of health-related quality of life (HRQL) | 5 minutes
  HRQL was measured by the Peds-QL 4.0 11,22. The 23-item Peds-QL 4.0 generic core scales encompass (a) physical functioning (eight items), (b) emotional functioning (five items), (c) social functioning (five items), and (d) school functioning (five items). The physical health summary score (eight items) is the same as the physical functioning scale. To create the psychosocial health summary score (15 items), the mean is computed as the sum of the items divided by the number of items answered in the emotional, social, and school functioning scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams University, Cairo, Abbasia, Egypt

REFERENCES:
- [Derived] El Samahy MH, Salah NY, Abdeen MS, Falastin BRK. Psychosocial aspects of continuous subcutaneous insulin infusion in children with type 1 diabetes in Egypt; a limited resources country perspective. Diabetol Metab Syndr. 2022 Jun 11;14(1):82. doi: 10.1186/s13098-022-00853-6. PMID 35690827